CLINICAL TRIAL: NCT02930031
Title: Evidence of a Redox-dependent Regulation of Immune Responses to Exercise-Induced Inflammation
Brief Title: Redox Status and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandra Sakelliou, PhD candidate in Department of Diabetes and Metabolism Unit, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NACEXERCISE2016
Record Dates: First submitted 2016-10-04; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Skeletal Muscle Damage; Aseptic Inflammation; Skeletal Muscle Function
Keywords: muscle injury; exercise; redox status; immune cells
MeSH Terms: conditions — Motor Activity | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-acetylcysteine (Experimental): orally in three daily dosages, at 20 mg/kg/day, daily for eight days after exercise
  Interventions: Dietary Supplement: n-acetylcysteine
- Placebo (Active Comparator): orally in three daily dosages, content: 500 mL drink that contained water (375 mL), sugar-free cordial (125 ml), and 2 g of low-calorie glucose/dextrose powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-acetylcysteine — 20 mg//kg/day, orally, daily for eight days following exercise
  Other Names: NAC
  Arms: n-acetylcysteine
Dietary Supplement: Placebo — 500 mL orally, daily for eight days following exercise
  Arms: Placebo

SUMMARY:
In this investigation the investigators utilized N-acetylcysteine (NAC) supplementation to enhance reduced glutathione (GSH) stores during an 8-day recovery period from a strenuous eccentric exercise protocol in order to test the hypotheses: i) redox status perturbations in skeletal muscle are pivotal for the immune responses and ii) antioxidant supplementation may alter immune cell responses following exercise-induced muscle microtrauma.

DETAILED DESCRIPTION:
The major thiol-disulfide couple of GSH and oxidized glutathione (GSSG) is a crucial regulator of the main transcriptional pathways regulating aseptic inflammation and recovery of skeletal muscle following aseptic injury. Antioxidant supplementation may hamper exercise-induced inflammatory responses.

The objective was to examine how thiol-based antioxidant supplementation affects immune mobilization following exercise-induced skeletal muscle microtrauma. In a two-trial, double-blind, crossover, repeated measures design, 10 young men received either placebo or NAC (20 mg/kg/day) immediately after a muscle-damaging exercise protocol (300 eccentric contractions) and for eight consecutive days. Blood sampling and performance assessment were performed pre-exercise, 2h post-exercise and daily for 8 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally trained (VO2max > 45 ml/kg/min)
* Engaged in regular exercise for ≥3 times/week for > 12 months
* non-smokers
* Abstain from exercise during the course of the two trials
* No consumption of performance-enhancing substances, antioxidants, caffeine, alcohol and/or medications during the study.

Exclusion Criteria:

* NAC intolerance
* Recent musculoskeletal injuries of the lower limbs
* Febrile illness
* History of muscle lesion.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in protein carbonyls in red blood cells | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Concentration of protein carbonyls
Changes in thiobarbituric acid reactive substances in red blood cells | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Thiobarbituric acid reactive substances concentration in red blood cells
Changes in total antioxidant capacity in serum | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
Changes in reduced glutathione in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Concentration of reduced glutathione in red blood cells
Changes in oxidized glutathione in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Concentration of oxidized glutathione in red blood cells
Changes in catalase activity in red blood cells | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
Changes in creatine kinase activity in serum | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
Changes in high sensitivity C-reactive protein in serum | Pre-exercise, 2 hours post-exercise, 1 day post-exercise, 2 days post-exercise, 3 days post-exercise
Changes in white blood cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
Changes in adhesion molecule concentration in blood | Pre-exercise, 2 hours post-exercise, 1 day post-exercise, 2 days post-exercise, 3 days post-exercise
  Measurement of soluble vascular cell adhesion molecule-1 (sVCAM-1) and soluble intercellular cell adhesion molecule-1 (sICAM-1) concentrations in plasma
Changes in cytokine concentration in serum | Pre-exercise, 2 hours post-exercise, 1 day post-exercise, 2 days post-exercise, 3 days post-exercise, 8 days post-exercise
  Measurement of interleukin-1β (IL-1β) and interleukin-6 (IL-6)
Changes in neutrophil count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of neutrophil count in blood
Changes in lymphocyte count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of lymphocyte count in blood
Changes in monocyte count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of monocyte count in blood
Changes in basophil count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of baseophil count in blood
Changes in eosinophil count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of eosinophil count in blood
Changes in T-helper cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of T-helper cell count in blood
Changes in T cytotoxic cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of T cytotoxic cell count in blood
Changes in natural killer-T (NK-T) cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of NK-T cell count in blood
Changes in 62L macrophage count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of 62L macrophage count in blood
Changes in B lympho cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of B lympho cell count in blood
Changes in natural killer (NK) cell count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of natural killer cell count in blood
Changes in macrophage count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of macrophage count in blood
Changes in HLA+/Macr+ macrophage count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of HLA+/Macr+ count in blood
Changes in 11B+ macrophage count in blood | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Cytofluorometric analysis of 11B+ macrophage count in blood

SECONDARY OUTCOMES:
Changes in muscle performance | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Assessment of maximal knee extensor eccentric peak torque on an isokinetic dynamometer at 60o/s.
Changes in delayed onset of muscle soreness | Pre-exercise, 2 hours post-exercise, daily for 8 consecutive days post-exercise
  Assessment of the delayed onset of muscle soreness by palpation of the vastus lateralis and rectus femoris following a squat motion
Maximal aerobic capacity | One day before exercise
  Assessment of maximal oxygen consumption
Body composition | One day before exercise
  Measurement of body composition by Dual Emission X-ray Absorptiometry (DXA)
Changes in dietary intake profile | One day before exercise and daily for 8 consecutive days post-exercise
  Assessment of dietary intake with emphasis on antioxidant element intake

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Mitrakou, Associate Prof., Study Director — Department of Diabetes and Metabolism Unit of the Department of Clinical Therapeutics, National and Kapodistrian University of Athens
Locations (1):
- University of Athens, Medical School, Department of Clinical Therapeutics, Athens, Greece